CLINICAL TRIAL: NCT07306429
Title: Evaluation of the Efficiency of Bone Born Intra Oral Distractor for Closure of Wide Alveolar Cleft
Acronym: BBID-WAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Hanaa Elmorsy, Assistant Lecturer at Oral and Maxillofacial Surgery department at AlAzhar University, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORSUR-10
Record Dates: First submitted 2025-11-30; First posted 2025-12-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Cleft; Distraction of Bone
Keywords: Alveolar Cleft; Bone Distraction
MeSH Terms: conditions — Diastasis, Bone

STUDY DESIGN:
Intervention Model Description: stereographic models were used for construction of bone-borne custom-made intraoral distractor
Masking Description: This wasn't applicable during surgery and follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone-Borne Intra-oral distractor (Experimental): Surgeries to fix the device were conducted under GA. Then latency period of seven days was applied. Activation was 0.5 mm twice a day. The transport segment touched the docking site then the Consolidation period is achieved. Follow up for 6 months.
  Interventions: Device: Bone-borne Intra oral distractor

INTERVENTIONS:
Device: Bone-borne Intra oral distractor — Evaluation of the efficiency of the Bone-Borne Intraoral distractors on wide Alveolar cleft

SUMMARY:
The study aimed to determine efficiency of Bone-Born Intraoral Distractor on wide Alveolar cleft patients

DETAILED DESCRIPTION:
Stereographic models were used for construction of bone-born custom-made intraoral distractor according to the inclusion and exclusion criteria, followed up to measure and determine the efficiency of the distractor

ELIGIBILITY:
Inclusion Criteria:

* Patients with wide alveolar clefts more than 8ml either unilateral or bilateral or median facial cleft.
* Patients who had previous failed grafting also may be included.
* Age range of patients 7-20 years old, with no gender prediction, able to read and sign the informed consent (parents)
* Patients with median facial clefts.

Exclusion Criteria:

* Narrow alveolar cleft
* Syndromic patients.
* Oral soft tissues defects, inflammation, infections and bone metabolism disturbance.
* Allergy to titanium implant.
* Patient with systemic disease and immunocompromised patient.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in alveolar cleft defect area measured by cone-beam computed tomography (CBCT) (minimum value: 0 mm²; no predefined maximum value; lower values indicate better outcome) | 6 months postoperative follow up
  The alveolar cleft defect area will be quantitatively measured using cone-beam computed tomography (CBCT). Preoperative and postoperative CBCT scans will be superimposed to calculate the change in defect area following distraction osteogenesis.
Change in tooth mobility assessed using Miller's Tooth Mobility Index (minimum score: 0; maximum score: 3; higher scores indicate worse mobility) | 6 months postoperative follow up
  Tooth mobility will be clinically evaluated using Miller's Tooth Mobility Index to detect and grade the degree of mobility before and after treatment.
Vitality of the transported bone segment assessed by clinical vitality indicators after transport distraction osteogenesis (binary outcome: viable / non-viable; viable outcome indicates better result) | 6 months follow up
  Vitality of the transported disk after transport distraction osteogenesis is measured through clinical indicators as No infection, No pain or inflammation, Stable transported segment, Successful consolidation phase.

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Elmorsy, Assis.Lec, Study Chair — Assistant lecturer of OMFs department Azhar University; Susan H Abdel Hakim, professor, Study Director — Professor of OMFs department azhar university; Wael Shawkat, Consultant, Study Director — Head of the department at the Health Insurance Hospital; Fatema khalifa, Assist.Prof, Study Director — Assistant Professor of OMFs Azhar university
Locations (1):
- Faculty of oral and dental medicine for Girls AlAzhar University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Detailed Protocol